CLINICAL TRIAL: NCT06598228
Title: Acute Kidney Injury and Recovery Mode in Pediatric Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Wei Gao, Head of the pediatric organ transplant unit, Tianjin First Central Hospital
Other Study IDs: 20240903-1
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Acute Kidney Injury; Pediatric Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- the group without acute kidney injury: Patients not diagnosed with acute kidney injury according to KDIGO(Kidney Disease: Improving Global Outcomes) criteria
  Interventions: Other: No Intervention: Observational Cohort
- the group with transient acute kidney injury: Patients diagnosed with acute kidney injury according to KDIGO(Kidney Disease: Improving Global Outcomes) criteria and recovered within 48h
  Interventions: Other: No Intervention: Observational Cohort
- the group with persistent acute kidney injury: Patients diagnosed with acute kidney injury according to KDIGO(Kidney Disease: Improving Global Outcomes) criteria and sustained over 48h
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — no intervention

SUMMARY:
Acute kidney injury (AKI) is a common complication after pediatric liver transplantation (PLT), and renal impairment after LT has proven to be related with increased graft failure and mortality. The recovery mode of kidney injury after PLT has not been systematically studied. Therefore, in this study the investigators aimed to systematically evaluate prognosis of AKI after PLT, combine the recovery mode of AKI with related risk factors, and establish a relationship between AKI and CKD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a liver transplant for the first time.
* Patients who were younger than 18 years of age at the time of transplant.

Exclusion Criteria:

* Patients with incomplete clinical data.
* Patients with less than 5 years of follow-up.
* Patients who have combined multiple solid organ transplants.
* Patients with preoperative renal impairment (eGFR<60ml/min/1.73 m2 or prior renal replacement therapy).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study was conducted on pediatric patients (aged ≤18 years) who received liver transplantation at Tianjin First Central Hospital in China between January 1, 2014 and December 31, 2018
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Graft survival | Based on the most recent follow-up before December 31, 2023. The investigators collected clinical data of patients from 2014 to 2018, and followed enrolled participants until at least 5 years after surgery
  Loss of graft is defined as patient death or secondary transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin First Central Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No